CLINICAL TRIAL: NCT03875742
Title: Interfascial Blocks Executed by Novice Operators in a Simulator Model: a Comparison of Two Types of Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019/SIMULARTI/ADC
Record Dates: First submitted 2019-02-22; First posted 2019-03-15 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia
Keywords: simulation; interfascial blocks; TAP block; needles

STUDY DESIGN:
Intervention Model Description: 70 anesthesia residents with low experience in interfascial blocks ( less than 15 interfascial blocks)will be asked to execute a Trasversus Abdominis Plane Block on "Trasversus Abdominis Plane Block Ultrasound Training Model" (BluePhantom) two times and they will be randomized in two groups.
  First group will execute the first Trasversus Abdominis Plane Block using UltraPlex 360(Braun) and the second Trasversus Abdominis Plane Block using STIMUPLEX D SH, 30°(Braun).
  Second group will execute the first Trasversus Abdominis Plane Block using STIMUPLEX D SH, 30°(Braun) and the second Trasversus Abdominis Plane Block using Ultraplex(Braun).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Ultraplex 360" (Other): This group will execute the first TAP block using "Ultraplex 360" (Braun) and the second TAP block using " STIMUPLEX D SH, 30°" (Braun)
  Interventions: Device: Ultraplex 360(Braun)
- " STIMUPLEX D SH, 30°" (Other): This group will execute the first TAP block using " STIMUPLEX D SH, 30°" (Braun) and the second TAP block using "Ultraplex 360" (Braun)
  Interventions: Device: STIMUPLEX D SH, 30°(Braun)

INTERVENTIONS:
Device: Ultraplex 360(Braun) — This group will use as first needle the "ultraplex 360" (Braun)
  Arms: "Ultraplex 360"
Device: STIMUPLEX D SH, 30°(Braun) — This group will use as first needle the " STIMUPLEX D SH, 30°" (Braun)
  Arms: " STIMUPLEX D SH, 30°"

SUMMARY:
This study will compare two different needles for interfascial blocks. All participants will execute the block on simulator with both needles. The participants will be randomized in two groups to choose the starting needle.

DETAILED DESCRIPTION:
Interfascial blocks are an emerging field of anesthesia. They are executed injecting local anesthetics inside a fascia plane using a needle.

Actually no evidence supports the use of a needle upon one other. Investigators would like to compare "Ultraplex 360®" (Braun) needle with " STIMUPLEX D SH, 30°"(Braun) while performing a Trasversus Abdominis Plane Block on BluePhantom simulator.

Ultraplex 360® (Braun) has an innovative surface pattern and clear coating that could result in better ultrasound visualization and tip identification.

ELIGIBILITY:
Inclusion Criteria:

* Novice interfascial block operators (< 15 interfascial blocks executed)
* informed consent

Exclusion Criteria:

* Exper Interfascial blocks operators

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Time to correct block execution | baseline
  Investigators will measure time needed to correctly perform the block in seconds. The chronometer will be started when the participant takes the ultrasound probe and will be stopped when 10 ml saline has been fully injected.

SECONDARY OUTCOMES:
Needle tip visualization | baseline
  Procedure will be recorded as a clip in ultrasound machine. Investigators will evaluate the time(seconds) during the procedure with a clear tip visualization. This time will be divided per total procedure time.
Participant Overall Satisfaction | baseline
  Participants satisfaction with the needle will be evaluated on a 0 to 10 scale at the end of the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Undecided